CLINICAL TRIAL: NCT00002639
Title: ANALYSIS OF THE EFFICACY OF SURAMIN IN RECURRENT MALIGNANT PRIMARY BRAIN TUMORS
Brief Title: Suramin in Treating Patients With Recurrent Primary Brain Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000064118; EUC-DON-9420; NCI-T94-0033O
Record Dates: First submitted 1999-11-01; First posted 2004-05-26 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2001-02

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult mixed glioma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Astrocytoma; Oligodendroglioma; Glioma; Gliosarcoma | interventions — Drug Therapy; Suramin

INTERVENTIONS:
Drug: chemotherapy
Drug: suramin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of suramin in treating patients with recurrent primary brain tumors following radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Estimate the efficacy of suramin in patients with recurrent primary brain tumors as measured by radiographic response, time to progression, and survival. II. Assess the toxic effects of suramin in this patient population.

OUTLINE: Single-Agent Chemotherapy. Suramin, SUR, NSC-34936.

PROJECTED ACCRUAL: If at least 1 of the first 14 patients experiences at least a partial response, a total of 25 patients will be entered over approximately 30 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Recurrent brain tumor based on one of the following: Tissue diagnosis if there was a prior diagnosis of astrocytoma or oligodendroglioma or if there is a question of radiation necrosis from prior interstitial brachytherapy Metabolic activity in excess of normal cortex measured by 18-fluorodeoxyglucose uptake on PET One of the following histologic types required: Glioblastoma multiforme Anaplastic astrocytoma Anaplastic oligodendroglioma Anaplastic mixed glioma Tumor progression required, i.e.: 28% increase in contrast-enhancing area or 50% increase in contrast- enhancing volume over at least 4 weeks Measurable disease required No history, surgical findings, or radiographic signs of intratumoral hemorrhage

PATIENT CHARACTERISTICS: Age: Over 15 Performance status: Karnofsky 50%-100% Life expectancy: At least 12 weeks Hematopoietic: WBC at least 3,000 Platelets at least 75,000 Hepatic: Bilirubin less than 1.5 mg/dL AST/ALT less than 3 times normal No history of bleeding disorder No hepatic disease resulting in hospitalization Renal: Creatinine less than 1.5 mg/dL No renal disease resulting in hospitalization Cardiovascular: No ongoing anticoagulation for deep vein thrombosis (DVT) No residual symptoms from DVT after discontinuation of anticoagulation No cardiac disease resulting in hospitalization Pulmonary: No pulmonary disease resulting in hospitalization Other: No peripheral neuropathy of any etiology HIV negative No pregnant or nursing women Adequate contraception required during and for 12 months following protocol therapy

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy for glioblastoma multiforme No more than 1 prior chemotherapy regimen for anaplastic astrocytoma, malignant oligodendroglioma, or malignant mixed glioma At least 4 weeks since chemotherapy (6 weeks since nitrosoureas or mitomycin) Endocrine therapy: Not specified Radiotherapy: Completion of 1 course of conventional external radiotherapy required At least 4 weeks since radiotherapy Surgery: Decompressive surgery for clinically suspected increased intracranial pressure performed prior to entry

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1995-07; Study Completion 2004-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey J. Olson, MD, Study Chair — Emory University
Locations (1):
- Department of Neurosurgery - Emory, Atlanta, Georgia, United States